CLINICAL TRIAL: NCT02094118
Title: Point-of-Care RBC Washing to Prevent Transfusion-Related Pulmonary Complications
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Duke University (Other); Vitalant Research Institute (Other)
Responsible Party: Principal Investigator, Daryl J. Kor, M.D., Associate Professor of Anesthsiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-005965
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-02

CONDITIONS: Blood Transfusion Complications
Keywords: Transfusion; RBC; cardiac; surgery; transfusion related acute lung injury (TRALI); transfusion associated circulatory overload (TACO)
MeSH Terms: conditions — Transfusion Reaction; Transfusion-Related Acute Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of care red blood cell transfusion (Active Comparator): Red blood cells that are administered in the normal fashion.
  Interventions: Biological: Standard of care red blood cell transfusion.
- Point-of-Care washed red blood cell transfusion (Experimental): Red blood cells that are washed at the point-of-care.
  Interventions: Biological: Point-of-care washed red blood cell transfusion.

INTERVENTIONS:
Biological: Point-of-care washed red blood cell transfusion.
  Arms: Point-of-Care washed red blood cell transfusion
Biological: Standard of care red blood cell transfusion.
  Arms: Standard of care red blood cell transfusion

SUMMARY:
This study is designed to determine if point-of-care washing of allogeneic Leukocyte-Reduced Red Blood Cells reduces pulmonary complications when compared to standard-of-care Leukocyte-Reduced Red Blood Cells in a cardiac surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years of age.
* Scheduled to have cardiac bypass surgery at Mayo Clinic in Rochester, Minnesota or Duke University Medical Center in Durham, North Carolina
* At risk for needing at least 4 units of blood during/after surgery

Exclusion Criteria:

* Emergency surgery
* Immunoglobulin A (IgA) deficiency
* History of severe recurrent transfusion reactions
* Refusal to receive allogeneic blood products
* Refusal to provide informed consent
* Prevalent lung injury prior to randomization
* Prevalent congestive heart failure prior to randomization
* Expected hospital stay < 48 hours
* Not anticipated to survive > 48 hours
* Previously enrolled in this trial
* No plan for placement of a pulmonary artery catheter
* Use of home oxygen therapy
* Complex RBC antibody profiles
* Need for the use of irradiated RBCs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2016-01; Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Kor, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warner MA, Welsby IJ, Norris PJ, Silliman CC, Armour S, Wittwer ED, Santrach PJ, Meade LA, Liedl LM, Nieuwenkamp CM, Douthit B, van Buskirk CM, Schulte PJ, Carter RE, Kor DJ. Point-of-care washing of allogeneic red blood cells for the prevention of transfusion-related respiratory complications (WAR-PRC): a protocol for a multicenter randomised clinical trial in patients undergoing cardiac surgery. BMJ Open. 2017 Aug 18;7(8):e016398. doi: 10.1136/bmjopen-2017-016398. PMID 28821525
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Red Blood Cell Transfusion: Red blood cells that are administered as standard of care.
  Standard of care red blood cell transfusion.
- Point-of-Care Washed Red Blood Cell Transfusion: Red blood cells that are washed at the point-of-care.
  Point-of-care washed red blood cell transfusion.
Period: Overall Study
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Started | 85 | 86
Completed | 73 | 81
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Red Blood Cell Transfusion: Red blood cells that are administered in the normal fashion.
  Standard of care red blood cell transfusion.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (11.4) | 65.0 (12.1) | 65.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 41 | 84
  Male | 42 | 45 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 81 | 78 | 159
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 15 | 29
  White | 66 | 64 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 85 | 86 | 171

OUTCOME MEASURES:

1. Primary Outcome: Biomarkers Associated With Transfusion-Related Acute Lung Injury and Transfusion Associated Circulatory Overload.
Description: This panel of biomarkers measures inflammation, altered coagulation, and endothelial activation all of which play key roles in the pathogenesis of lung injury.
Time Frame: 18 hours after the initiation of the first red blood cell transfusion.
Population: Patients undergoing cardiac surgery who were predicted to be at high risk for requiring red blood cell transfusion.
Measure: Median (Inter-Quartile Range); unit: units on a scale (pg/ml)
Groups:
- Standard of Care Red Blood Cell Transfusion: Red blood cells transfusion that were administered in the standard of care
- Point-of-Care Washed Red Blood Cell Transfusion: Red blood cells transfusion that were washed at the point-of-care.
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (pg/ml)
  IL-6 | 101 [57 to 197] | 105 [70 to 191]
  IL-8 | 12 [6 to 23] | 15 [7 to 26]
  vWF | 107 [84 to 137] | 111 [74 to 142]
  RAGE | 3262 [2326 to 6899] | 4516 [2354 to 5907]
  SP_D | 7238 [4962 to 11900] | 7061 [4470 to 13318]
  PAI_1 | 73418 [38900 to 196491] | 53829 [21044 to 151009]
  ICAM_1 | 404914 [313796 to 513060] | 404129 [309411 to 538055]

2. Primary Outcome: Number of "Off-protocol" Transfusions
Description: The number of standard issued red blood cell units that were transfused to study participants in the washed red blood cell arm of the trial. Additionally, emergency red blood cell transfusions in the standard issued arm of the trial that were administered outside of the study protocol were also included to the definition of "off protocol" transfusion.
Time Frame: Day of surgery. Approximately 1 day.
Measure: Number; unit: transfusions
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
transfusions | 3 | 22

3. Primary Outcome: Change in Recipient Hemoglobin
Description: Change in Hemoglobin from pre-transfusion to post-transfusion
Time Frame: Pre to 6 hours post transfusion
Measure: Median (Inter-Quartile Range); unit: units on a scale (g/dl)
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (g/dl) | 2.6 [1.6 to 3.6] | 2.3 [1.4 to 3.1]

4. Primary Outcome: Change in Recipient Cell Free Hemoglobin(CFH)
Description: Change in CFH from pre-transfusion to worst (highest/maximum) post-transfusion
Time Frame: Pre transfusion until study day 5 or hospital discharge, approximately 5 days
Measure: Median (Inter-Quartile Range); unit: units on a scale (mg/dl)
Groups:
- Standard of Care Red Blood Cell Transfusion: Red blood cells that are administered as standard of care.
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (mg/dl) | 22.8 [8.9 to 52] | 23 [6.6 to 58.4]

5. Primary Outcome: Change in Haptoglobin
Description: Change in Haptoglobin from pre-transfusion to worst (minimum) post-transfusion
Time Frame: Pre transfusion to study day 5 or hospital discharge, approximately 5 days
Measure: Median (Inter-Quartile Range); unit: units on a scale (mg/dl)
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (mg/dl) | -48.5 [-95 to -16.5] | -54 [-103 to -7]

6. Secondary Outcome: Duration of Mechanical Ventilation
Description: Number of hours subject received mechanical ventilation.
Time Frame: Up to hospital day 28, or discharge, whichever comes first
Measure: Median (Inter-Quartile Range); unit: units on a scale (hours)
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (hours) | 10.3 [5.6 to 23.5] | 10.8 [5.6 to 20.1]

7. Secondary Outcome: Duration of Oxygen Supplementation
Description: Number of hours subjects received supplemental oxygen.
Time Frame: Up to day 28, or hospital discharge, whichever comes first
Measure: Median (Inter-Quartile Range); unit: units on a scale (hours)
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (hours) | 84.7 [45.5 to 142.7] | 89.5 [39.9 to 180.4]

8. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score
Description: Worst SOFA score between Day 1 and Day 5. SOFA scores range from 0-24 with 0 meaning no organ dysfunction and 24 means severe dysfunction of all organ systems evaluated. Each of 6 organ systems are scored on a 0-4 scale with the cumulative score being the total SOFA score.
Time Frame: Through postoperative day 5.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale | 12 [10 to 14] | 13 [11 to 14]

9. Secondary Outcome: Hospital Length of Stay
Description: Number of days subject remained in the hospital following their surgical procedure. If the number of days the subject remained in the hospital exceeded 28, a value of 28 is assigned.
Time Frame: Up to day 28
Measure: Median (Inter-Quartile Range); unit: units on a scale (days)
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
units on a scale (days) | 12 [9 to 17] | 12 [9 to 17]

10. Secondary Outcome: Post Transfusion Respiratory Complications.
Description: Development of transfusion-related lung injury (TRALI) or transfusion-associated circulatory overload (TACO).
Time Frame: Up to day 28
Measure: Number; unit: participants
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
Number analyzed (Participants) | 73 | 81
participants
  TACO | 7 | 5
  TRALI | 1 | 0

ADVERSE EVENTS:
Time Frame: From randomization to hospital discharge, death, or day 28 (whichever occurs first).
Arm/Group | Standard of Care Red Blood Cell Transfusion | Point-of-Care Washed Red Blood Cell Transfusion
All-Cause Mortality (participants affected / at risk) | 2/85 | 3/86
Serious Adverse Events (participants affected / at risk) | 0/85 | 7/86
Other Adverse Events (participants affected / at risk) | 0/85 | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Red Blood Cell Transfusion (N=85) | Point-of-Care Washed Red Blood Cell Transfusion (N=86)
hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Profound Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT02094118/Prot_SAP_000.pdf